CLINICAL TRIAL: NCT01568970
Title: Multidisciplinary Return-to-work Rehabilitation and Return-to-work Follow-up, a Randomized Study of Patients With Complex Symptom Disorders
Brief Title: Multidisciplinary Return-to-work Rehabilitation and Return-to Work Follow-up
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2010/2404
Record Dates: First submitted 2012-03-08; First posted 2012-04-02 (Estimated); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Complex Symptom Disorders
Keywords: rehabilitation; return to work; sick leave
MeSH Terms: interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Return to work follow-up (Experimental): Regular contact between the patient and his/her caretaker at the rehabilitation center over a 6 month period, including joint communication between patient, caretaker at the rehabilitation center and stake holders such as social security office, general practitioner and workplace.
  Interventions: Behavioral: Return-to-work Rehabilitation + Follow up
- Standard follow-up (Active Comparator): Standard follow-up of the patient after ended rehabilitation by the return-to-work stakeholders, ie. the general practitioner, social security office and the employer. Limited contact between the caretaker at the rehabilitation center and the patient and stakeholders.
  Interventions: Behavioral: Return-to-work rehabilitation

INTERVENTIONS:
Behavioral: Return-to-work Rehabilitation + Follow up — 3 1/2 weeks of Return-to-work rehabilitation followed by 6 months of Return-to-work follow-up
  Other Names: Acceptance commitment therapy
  Arms: Return to work follow-up
Behavioral: Return-to-work rehabilitation — 3 1/2 weeks of Return-to-work rehabilitation followed by standard follow-up
  Other Names: Acceptance commitment therapy
  Arms: Standard follow-up

SUMMARY:
The large number of people on long-term sick leave is a major public health concern in Norway. The main causes of disability are musculoskeletal and mental disorders. Long-term sick leave causes a decline in individual life-quality, is associated with increased risk for mental disorders and represents a very large cost for the Norwegian society.

The purpose of this study is to determine whether the patients included return to work after rehabilitation at Hysnes Rehabilitation Centre. This includes an investigation of what is considered to be the effect of Return-to-work rehabilitation measured before, during and after the stay at the rehabilitation centre:

The study specifically looks at the effect of structured and standardized return-to-work follow up of the patient, including contact with stakeholders (general practitioner, social security office and workplace).

In addition there is a need to describe the patients participating in the program. The aetiology of complex symptom disorders is poorly understood and the role of genetics and stress is not translatable to a complex symptom population. This complicates the transition from current biological research to a clinical use regarding these patients. If the investigators can assist in understanding how these patients, who are multiusers of health care and have received sickness benefit for a long time, develop their disorders and symptoms, it will be of great importance to the Norwegian community. Therefore the study consists of multimodal measurements of the patients before, during and after a rehabilitation programme at Hysnes Rehabilitation Centre. These measures include genotype, saliva cortisol, medical-, psychological-, physiological diagnostics and work related factors.

Related aims:

Investigate if multidisciplinary treatment based on acceptance and commitment therapy, contributes to normalisation of cortisol release with regards to a standardized stress test.

See wether individual differences regarding the stress profile can predict return to work in patients with complex symptom disorders.

Investigate genetic risk factors in relation to Return to Work rehabilitation and identify treatment moderators in a multidisciplinary rehabilitation program.

ELIGIBILITY:
Inclusion criteria:

* Age between 18-59 years
* A self defined goal of increasing their work ability and work participation within a period of no more than six months
* They fill the criteria of a complex symptom disorder, or they are diagnosed with a common mental disorder
* A satisfactory level of examination and treatment to participate at Hysnes Rehabilitation Centre
* Sick leave > 8weeks or receiving work ability assessment benefit for any diagnosis, except as stated below.
* On a level of linguistic, physical and mental function required to participate in the rehabilitation

Exclusion criteria:

* Ongoing alcohol/drug abuse
* Ongoing psychosis, ongoing manic episode or suicide risk
* Pregnancy

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 214 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Return to work | 1 year after the end of the stay at the rehabilitation center.
  Differences in cumulative days of sick leave, as reported by the government database "FD-Trygd".

SECONDARY OUTCOMES:
quality of life | 5 years after the end of the rehabilitation stay
  Quality of life is assessed by 15D, SF8 and function subscale in SF-36
Functional status | 5 year after the end of the rehabilitation stay
  Functional status will be measured with elements from the Norwegian Function Assessment Scale (Osteras et al., 2007) and the function subscale of SF-36 (Ware Jr & Sherbourne, 1992)
level of symptoms (somatic and psychological) | 5 year after the end of the rehabilitation stay,
  The Hospital Anxiety and Depression Scale (HADS) measure changes in anxiety and depression.
  Changes regarding physical and mental fatigue are registered through the Chalder Fatigue Questionnaire.
  Changes in participants subjective experience of pain measured by numerical rating scale (NRS)

CONTACTS AND LOCATIONS:
Overall Officials: Petter Borchgrevink, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Hysnes Helsefort, St Olavs Hospital, Trondheim, Norway

REFERENCES:
- [Result] Hara KW, Bjorngaard JH, Brage S, Borchgrevink PC, Halsteinli V, Stiles TC, Johnsen R, Woodhouse A. Randomized Controlled Trial of Adding Telephone Follow-Up to an Occupational Rehabilitation Program to Increase Work Participation. J Occup Rehabil. 2018 Jun;28(2):265-278. doi: 10.1007/s10926-017-9711-4. PMID 28597308
- [Derived] Vethe D, Kallestad H, Jacobsen HB, Landro NI, Borchgrevink PC, Stiles TC. The Relationship Between Improvement in Insomnia Severity and Long-Term Outcomes in the Treatment of Chronic Fatigue. Front Psychol. 2018 Sep 21;9:1764. doi: 10.3389/fpsyg.2018.01764. eCollection 2018. PMID 30298037